CLINICAL TRIAL: NCT05547776
Title: Mindfulness-Based Stress Reduction App for African American Caregivers of People With Chronic Conditions
Brief Title: Mindfulness Based Stress Reduction App for African American Caregivers (MBSR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: COG Analytics (Other)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R41AG071168-01A1 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: This is a feasibility trial with a single group of 30 participants who are using an app and providing feedback on the app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms and Interventions (Experimental): Mindfulness App Use
  Participants will have the opportunity to use the mindfulness app for four weeks.
  Interventions: Behavioral: Mindfulness app

INTERVENTIONS:
Behavioral: Mindfulness app — The mindfulness app contains 6 modules with a variety of features to help caregivers reduce their stress.

SUMMARY:
The study investigators are developing and testing a mobile-friendly web-based app that contains features related to mindfulness and reducing stress for African American informal caregivers of people with chronic conditions. The purpose of the app is to help a vulnerable population reduce stress by learning and practicing mindfulness activities.

DETAILED DESCRIPTION:
For Aim 1, the study investigators conducted 10 formative interviews with African American caregivers and key informants to elicit recommendations for features to be included in the app as well as feedback on preliminary ideas for features. For Aim 2, the study investigators developed the programming for the app with the desired features, which included modules for journaling, tracking stress ratings, practicing mindfulness exercises by using two videos and two audio tracks developed for the app, and viewing weekly suggestions for caregiver/care recipient bonding activities, inspirational quotes and positive affirmations. For Aim 3, the study investigators are testing the app using a feasibility trial with 30 caregiver participants. The study participants answer questions on depression, anxiety, perceived stress, overload and self-compassion at baseline and follow-up. Participants are instructed to use the app for four weeks and to return for their follow-up visit to fill out the same surveys assessed at baseline plus a satisfaction questionnaire to assess their evaluation of the app. These data will inform future enhancements, which will be proposed in a Phase II SBIR/STTR application.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver participants will be screened for the ability to speak English. In addition, the caregivers must currently be providing support for a person living with HIV. Support can include: 1) emotional support, 2) physical support, 3) financial support, 4) opportunities for social participation, and/or 5) health advice.

Exclusion Criteria:

* Psychiatric problems such as untreated psychosis, which could preclude their ability to successfully adhere to the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | 4 weeks
  Perceived stress scores entered into the app by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Mitchell, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
None formulated.